CLINICAL TRIAL: NCT07147153
Title: Investigation of the Relationship Between Functional Capacity, Sleep Quality, and Cognitive Functions in Individuals With Obesity Hypoventilation Syndrome
Brief Title: Functional Capacity, Sleep Quality, and Cognitive Function in Obesity Hypoventilation Syndrome
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Sponsor
Other Study IDs: E-29624016-050.99-3179056
Record Dates: First submitted 2025-08-19; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Obesity Hypoventilation Syndrome (OHS)
Keywords: obesity; hypoventilation syndrome; cognitive functions
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group ı: Individuals diagnosed with Obesity Hypoventilation Syndrome by a pulmonologist based on polysomnography results.
- Group II: Individuals with simple obesity (BMI >30 kg/m²), comparable to Group 1 in terms of age and sex, who had an Apnea-Hypopnea Index (AHI) <5 on polysomnography or a STOP-Bang score <3.

SUMMARY:
Introduction:

Obesity Hypoventilation Syndrome (OHS) is defined as the coexistence of obesity (BMI ≥ 30 kg/m²), daytime hypercapnia (PaCO₂ > 45 mmHg) in the absence of other causes of hypoventilation, and sleep-disordered breathing. OHS represents the most severe form of obesity-related respiratory failure and leads to serious consequences such as increased mortality rates, chronic heart failure, pulmonary hypertension, and hospitalisations due to acute or chronic hypercapnic respiratory failure.

Aim:

The aim of this study is to evaluate cognitive functions in individuals with OHS and to investigate the relationship between cognitive functions, sleep quality, and functional capacity. A review of the literature indicates that cognitive functions in OHS have not been sufficiently examined, and existing studies mainly focus on cognitive impairment in individuals with obstructive sleep apnea syndrome (OSAS). However, OHS may also cause cognitive deficits, and therefore, patients should be assessed from this perspective. Cognitive impairment may negatively affect participation in pulmonary rehabilitation programs and reduce the benefits gained from such programs. Moreover, psychological conditions such as depression and anxiety may also influence the success of pulmonary rehabilitation. Thus, identifying cognitive impairment and its association with parameters such as functional capacity and sleep quality is of great importance. Early detection of cognitive deficits may provide positive outcomes for both patients and the healthcare system.

Methods:

The study will include 18 individuals with OHS diagnosed by a pulmonologist through polysomnographic evaluation at the Department of Pulmonology, Istanbul University, Istanbul Faculty of Medicine, along with 18 age- and sex-matched individuals with simple obesity (BMI >30 kg/m²). All participants will be evaluated at the Department of Pulmonology, Istanbul University, Istanbul Faculty of Medicine. Body composition will be assessed using bioelectrical impedance analysis with the "Tanita BC-545N Body Composition Monitor." Functional exercise capacity will be evaluated with the Incremental Shuttle Walk Test (ISWT) and the Six-Minute Walk Test (6MWT). Cognitive functions and attention will be assessed using the Montreal Cognitive Assessment (MoCA) and the Visual Reaction Time Test. Daytime sleepiness will be measured with the Epworth Sleepiness Scale (ESS), while sleep quality will be evaluated with the Pittsburgh Sleep Quality Index (PSQI). Psychological status will be assessed using the Depression Anxiety Stress Scale (DASS-21).

Statistical analyses will be conducted using the Statistical Package for Social Sciences (SPSS, version 21.0). Arithmetic mean, standard deviation (SD), and confidence intervals (CI) will be presented in tables and figures. The Shapiro-Wilk test will be applied to assess the normality of data distribution. For comparisons between the OHS and simple obesity groups, the Independent Samples T-Test will be used for normally distributed data, while the Mann-Whitney U test will be used for non-normally distributed data. Pearson or Spearman correlation analyses will be performed to investigate the relationship between functional capacity, sleep quality, and cognitive functions.

DETAILED DESCRIPTION:
Obesity Hypoventilation Syndrome (OHS) is defined as the combination of obesity (BMI ≥ 30 kg/m²), daytime hypercapnia (PaCO₂ > 45 mmHg) in the absence of other pathologies causing hypoventilation, and sleep-disordered breathing. OHS represents the most severe form of obesity-related respiratory failure and is associated with serious consequences, including increased mortality rates, chronic heart failure, pulmonary hypertension, and hospitalizations due to acute-on-chronic hypercapnic respiratory failure. The pathophysiology of OHS is multifactorial. Factors include reduced lung compliance; decreased lung volumes resulting from impaired respiratory mechanics; increased CO₂ production and respiratory workload; and hormonal influences such as decreased leptin and insulin-like growth factor-1 (IGF-I) levels. Reduced lung compliance and increased airway resistance lead to a higher respiratory workload, which contributes to respiratory muscle fatigue. Impaired respiratory mechanics and reduced respiratory muscle strength result in diminished functional capacity.

Sleep quality is known to be highly important for the maintenance of cognitive functions, and poor sleep quality is considered a risk factor for cognitive decline. In pulmonary diseases such as obstructive sleep apnea syndrome (OSAS), chronic obstructive pulmonary disease (COPD), and asthma, sleep quality is adversely affected for various reasons. Previous studies have reported that in these conditions-where sleep quality is compromised-cognitive functions are also impaired, with concurrent problems such as anxiety and depression, and that there is a correlation between disease severity and the degree of cognitive impairment. Cognitive impairment in these patients, especially marked cognitive decline, can negatively affect participation in pulmonary rehabilitation programs, self-management of treatment, adherence to medications/devices, and overall independence, thereby reducing the potential benefits of rehabilitation. Furthermore, psychological conditions such as depression and anxiety may also influence pulmonary rehabilitation outcomes, and it has been reported that identifying and managing these problems can enhance treatment efficacy. Components such as psychosocial support and patient education are considered important for minimizing the negative effects of cognitive or emotional factors on treatment outcomes.

In both OHS and OSAS, similar symptoms-including intermittent nocturnal hypoxemia, sleep fragmentation, excessive daytime sleepiness, and snoring-negatively affect sleep quality, increase daytime somnolence, and reduce quality of life. While sleep quality is impacted in both disorders due to similar pathophysiological mechanisms, numerous studies have examined the role of OSAS or obesity in cognitive functions and psychiatric disorders, yet no studies have been found that specifically investigate cognitive functions in patients with OHS. It has been suggested that intermittent hypoxia and hypercapnia in OHS may lead to cognitive impairment; however, sufficient clinical evidence to support this is lacking.

This study aims to assess cognitive functions in individuals with OHS and to investigate the relationship between cognitive functions, sleep quality, and functional capacity. A review of the literature reveals that cognitive functions in OHS have not been sufficiently examined, with most studies focusing on cognitive status in individuals with OSAS. Nevertheless, OHS may also cause cognitive impairment, and individuals should be evaluated from this perspective. Cognitive impairment in patients can adversely affect participation in pulmonary rehabilitation programs and the benefits gained from such interventions. Additionally, psychological factors such as depression and anxiety can also influence pulmonary rehabilitation outcomes. Therefore, identifying cognitive impairment and clarifying its relationship with parameters such as functional capacity and sleep quality is of considerable importance. Early detection of cognitive impairment in these individuals could provide positive feedback for both patients and the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Diagnosed with OHS by a pulmonologist
* For individuals with simple obesity: BMI between 30 and 40 kg/m², Apnea-Hypopnea Index (AHI) < 5 on polysomnography, or STOP-Bang score < 3
* Ability to communicate in written and spoken Turkish

Exclusion Criteria:

* Presence of any additional severe respiratory disease
* Presence of orthopedic, neurological, cardiovascular, or respiratory conditions preventing exercise testing
* For individuals with simple obesity: presence of OSAS risk factors such as severe snoring or witnessed apnea
* Presence of any psychological or psychiatric disorder that could affect cognitive functions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Obesity Hypoventilation Syndrome who applied to the Department of Pulmonary Diseases at Istanbul University Istanbul Faculty of Medicine, met the inclusion criteria for the study, and were diagnosed through polysomnographic evaluation by a Pulmonary Disease specialist.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Incremental Shuttle Walk Test (ISWT) | At baseline (immediately after informed consent)
  The ISWT is a field test consisting of 12 levels in which walking speed increases progressively. Participants are required to walk back and forth between two cones placed 10 meters apart, performing at their maximal capacity until symptom limitation. The test will be terminated if the patient is unable to maintain the required pace due to dyspnea, upon reaching maximal heart rate, or if the participant is more than 0.5 m behind the cone at the designated signal. The number of completed shuttles will be recorded, along with pre- and post-test measurements of blood pressure, heart rate, oxygen saturation, and dyspnea and leg fatigue scores using the Modified Borg Scale.
Montreal Cognitive Assessment (MoCA) | At baseline (immediately after informed consent)
  Cognitive functions including selective and sustained attention, information processing speed, short-term memory, and reaction time will be evaluated using standardized tests. To minimize environmental influences, all assessments will be conducted under identical conditions-in a quiet room with consistent physical settings-at the same time of day and by the same researchers for each participant.
  The MoCA will be used as a cognitive screening tool. It evaluates executive functions, attention and concentration, memory, language, abstract thinking, visuospatial skills, orientation, and calculation. The test takes approximately 10 minutes, and scores are calculated out of 30. A cutoff score of 26 is used; scores below this threshold indicate mild cognitive impairment.

SECONDARY OUTCOMES:
Six-Minute Walk Test (6MWT) | At baseline (immediately after informed consent)
  Submaximal functional exercise capacity will be assessed with the 6MWT following ATS guidelines (86). Participants will be instructed to walk at their own pace along a 30-meter flat corridor for six minutes, covering as much distance as possible. Before the test, participants will rest in a seated position for 10 minutes, after which baseline SpO₂, heart rate, blood pressure, and Modified Borg Scale scores for dyspnea and fatigue will be obtained. The same measurements will be repeated after the test. The six-minute walking distance (6MWD) will be recorded in meters.
Visual Reaction Time | At baseline (immediately after informed consent)
  Reaction time will be assessed using the Simple Visual Reaction Time Task implemented via Inquisit version 6.0, a computer-based software platform that also includes cognitive tests and games. In this test, participants are instructed to press the space bar as quickly as possible when a red circle appears at random intervals (2000-8000 ms) on a white screen. Two sets of 20 trials will be performed, and the average will be calculated. The fastest, slowest, and mean reaction times will be recorded as outcomes.
Epworth Sleepiness Scale (ESS) | At baseline (immediately after informed consent)
  The ESS consists of 8 items assessing the likelihood of dozing off during daily activities. Each item is scored from 0 (never) to 3 (always). A total score ≥10 indicates excessive daytime sleepiness. The Turkish validity and reliability of the scale have been established, with high internal consistency across the eight items (Cronbach's α = 0.80).
Pittsburgh Sleep Quality Index (PSQI) | At baseline (immediately after informed consent)
  The PSQI is a 24-item self-reported questionnaire that evaluates sleep quality and disturbances over the past month (25). Its Turkish version has demonstrated validity and reliability (26). The index consists of seven components-subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction-scored on a scale of 0-3. The sum of these component scores yields a global PSQI score ranging from 0 to 21, with scores >5 indicating poor sleep quality.
Depression Anxiety Stress Scale (DASS-21) | At baseline (immediately after informed consent)
  Psychological status will be evaluated using the Depression Anxiety Stress Scale (DASS-21). Originally developed by Lovibond & Lovibond (1995) as a 42-item scale, consisting of 14 items for depression, 14 for anxiety, and 14 for stress (27), the shortened 21-item version (DASS-21) was later developed by Henry & Crawford (2005). The Turkish validity and reliability of the DASS-21 were confirmed by Sarıçam. The scale consists of three subscales (depression, anxiety, and stress), each containing seven items, rated on a 4-point Likert scale (0 = never, 1 = sometimes, 2 = often, 3 = always). Higher total scores indicate greater severity of depression, anxiety, or stress. Reported Cronbach's alpha coefficients are α=0.87 for depression, α=0.85 for anxiety, and α=0.81 for stress. Test-retest reliability (ICC) has been reported as r=0.68 for depression, r=0.66 for anxiety, and r=0.61 for stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Argun Baris S, Tuncel D, Ozerdem C, Kutlu H, Onyilmaz T, Basyigit I, Boyaci H, Yildiz F. The effect of positive airway pressure therapy on neurocognitive functions, depression and anxiety in obesity hypoventilation syndrome. Multidiscip Respir Med. 2016 Oct 11;11:35. doi: 10.1186/s40248-016-0071-2. eCollection 2016. PMID 27766147
- [Result] Kielb SA, Ancoli-Israel S, Rebok GW, Spira AP. Cognition in obstructive sleep apnea-hypopnea syndrome (OSAS): current clinical knowledge and the impact of treatment. Neuromolecular Med. 2012 Sep;14(3):180-93. doi: 10.1007/s12017-012-8182-1. Epub 2012 May 9. PMID 22569877
- [Result] Ranzini L, Schiavi M, Pierobon A, Granata N, Giardini A. From Mild Cognitive Impairment (MCI) to Dementia in Chronic Obstructive Pulmonary Disease. Implications for Clinical Practice and Disease Management: A Mini-Review. Front Psychol. 2020 Feb 28;11:337. doi: 10.3389/fpsyg.2020.00337. eCollection 2020. PMID 32184750
- [Result] Pierobon A, Sini Bottelli E, Ranzini L, Bruschi C, Maestri R, Bertolotti G, Sommaruga M, Torlaschi V, Callegari S, Giardini A. COPD patients' self-reported adherence, psychosocial factors and mild cognitive impairment in pulmonary rehabilitation. Int J Chron Obstruct Pulmon Dis. 2017 Jul 18;12:2059-2067. doi: 10.2147/COPD.S133586. eCollection 2017. PMID 28790808
- [Result] Sharafkhaneh A, Giray N, Richardson P, Young T, Hirshkowitz M. Association of psychiatric disorders and sleep apnea in a large cohort. Sleep. 2005 Nov;28(11):1405-11. doi: 10.1093/sleep/28.11.1405. PMID 16335330
- [Result] Andreou G, Vlachos F, Makanikas K. Effects of chronic obstructive pulmonary disease and obstructive sleep apnea on cognitive functions: evidence for a common nature. Sleep Disord. 2014;2014:768210. doi: 10.1155/2014/768210. Epub 2014 Feb 6. PMID 24649370
- [Result] McNicholas WT, Hansson D, Schiza S, Grote L. Sleep in chronic respiratory disease: COPD and hypoventilation disorders. Eur Respir Rev. 2019 Sep 25;28(153):190064. doi: 10.1183/16000617.0064-2019. Print 2019 Sep 30. PMID 31554703
- [Result] Olaithe M, Bucks RS, Hillman DR, Eastwood PR. Cognitive deficits in obstructive sleep apnea: Insights from a meta-review and comparison with deficits observed in COPD, insomnia, and sleep deprivation. Sleep Med Rev. 2018 Apr;38:39-49. doi: 10.1016/j.smrv.2017.03.005. Epub 2017 Mar 30. PMID 28760549
- [Result] Spira AP, Chen-Edinboro LP, Wu MN, Yaffe K. Impact of sleep on the risk of cognitive decline and dementia. Curr Opin Psychiatry. 2014 Nov;27(6):478-83. doi: 10.1097/YCO.0000000000000106. PMID 25188896
- [Result] Dusgun ES, Aslan GK, Abanoz ES, Kiyan E. Respiratory Muscle Endurance in Obesity Hypoventilation Syndrome. Respir Care. 2022 May;67(5):526-533. doi: 10.4187/respcare.09338. Epub 2022 Mar 22. PMID 35318239
- [Result] Iftikhar IH, Roland J. Obesity Hypoventilation Syndrome. Clin Chest Med. 2018 Jun;39(2):427-436. doi: 10.1016/j.ccm.2018.01.006. PMID 29779600
- [Result] Mokhlesi B, Masa JF, Brozek JL, Gurubhagavatula I, Murphy PB, Piper AJ, Tulaimat A, Afshar M, Balachandran JS, Dweik RA, Grunstein RR, Hart N, Kaw R, Lorenzi-Filho G, Pamidi S, Patel BK, Patil SP, Pepin JL, Soghier I, Tamae Kakazu M, Teodorescu M. Evaluation and Management of Obesity Hypoventilation Syndrome. An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2019 Aug 1;200(3):e6-e24. doi: 10.1164/rccm.201905-1071ST. PMID 31368798